CLINICAL TRIAL: NCT02502214
Title: Feasibility Study of Preimplantation Genetic Diagnosis for Single-gene Disorders by Using Nextgeneration Sequencing
Brief Title: Feasibility Study of Preimplantation Genetic Diagnosis for Single-gene Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6195
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Preimplantation Diagnosis
Keywords: Preimplantation Genetic Diagnosis; PGD; Next-Generation Sequencing; NGS; Single-Gene disorders; Cystic Fibrosis; CFTR; Single-cell analysis; PCR; SNP; Whole Genome Amplification
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preimplantation Genetic Diagnosis (PGD) for monogenic diseases is usually performed by multiplex PCR combining polymorphic microsatellites familial analysis and, where possible, couple-specific mutation detection. Single-cell multiplex PCR developments are costly and time-consuming. We propose to test and clinically validate a targeted next-generation sequencing approach for the PGD for cystic fibrosis. This technique would allow a PGD for probably almost every couple asking for it in our centre, without a previous couple-specific development (but only a preliminary familial analysis). It will be based on haplotyping using a large number of SNPs and mutation detection. A clinical validation will be performed by reanalysing non-transferable embryos obtained after PGD for cystic fibrosis, with couple's informed consent. Concordance of the results between PGD and reanalysis by NGS will be achieved and if validated, this technique may be applied to future PGD for cystic fibrosis in our centre. The same technique may then be applied for other PGD indications for which a set-up is often needed.

ELIGIBILITY:
Inclusion Criteria:

* Age> or = 18 years
* Couples at risk of transmitting cystic fibrosis
* asking for a PGD in Strasbourg
* DNA samples available at the laboratory for:

  * The couple
  * A related with CFTR status known
  * Having signed an informed consent

Exclusion Criteria:

* Inability to give informed consent (understanding difficulties...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Preimplantation Diagnosis (DPI) may be offered to couples at risk of transmitting a serious genetic disease to their offspring
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-11-12 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Monogenic diseases | for the duration of hospital stay, up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire de Diagnostic préimplantatoire Site du CMCO, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No